CLINICAL TRIAL: NCT02509442
Title: Pilot Study: Measure of the Potential Evoked With Electroencephalography and Electrocorticography by Electric Stimulation of the Brain During the Neurosurgery Awakened of the Infiltrative Glioma of Low Grade (OMS Type II)
Brief Title: Measure of the Potential Evoked by Electric Stimulation
Acronym: PE&CE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: National Development and Research Institutes, Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 9530
Record Dates: First submitted 2015-04-22; First posted 2015-07-28 (Estimated); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Low Grade Glioma of Brain
Keywords: mapping brain functions; Direct electric stimulation (DES); potential evoked

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Diffusion of direct electric stimulation (Other): Neurosurgery awakened
  Interventions: Procedure: Diffusion of direct electric stimulation

INTERVENTIONS:
Procedure: Diffusion of direct electric stimulation — During the neurosurgery awakened consisting in resecting a low-rank infiltrative glioma , the potential evoked further to the direct electric stimulation of the brain will be recorded by electroencephalography and electrocorticography.
  Other Names: Neurosurgery awakened

SUMMARY:
This study is about an experimental biomedical monocentric search concerning twelves patients presenting a infiltrative glioma of low rank OMS type II and realizing a surgery awakened on the site of the CHU of Montpellier.

The objective of this search is to understand exactly how the electric impulses, delivered by the neurosurgeon to make a functional mapping of the brain during the surgery awakened by tumors infiltrates of low rank, propagate in this one and to identify the nervous networks inhibited by these electric impulses.

Having verified the eligibility of the patients and having obtained their consent, they will be included in the study. Before the beginning of the surgery, the electroencephalography activity of the brain of every patient will be recorded. Before and after the surgical resection, the electrocorticography activity will be recorded.

The collected data will then be analyzed, after the operation. Analyses will try to identify what we call potential evoked by the stimulation and which are small electric waves which appear after the electric stimulation was delivered.

DETAILED DESCRIPTION:
All the surgical operations will be realized by Professor Hugues DUFFAU. The DEMAR-INRIA team will assure the collection and the data processing electrophysiological, the management of the data and the methodological follow-up, as well as the writing of the report and the distribution of the results.

The quality assurance will be assured by a "minimal" monitoring by an assistant of clinical research for the department of the research and the innovation, to Montpellier, which will verify principally the consents.

The electrophysiological data digitized will be stored in the form of computer files via PowerLab.

All the analyses of treatment of signals required to highlight the potential evoked will be realized with the software Matlab.

ELIGIBILITY:
Inclusion Criteria:

* Patient carrier of a low-rank infiltrative glioma (OMS Type II) and presenting the indications to benefit from a surgical care in condition awakened for the first time.
* Patient capable of understanding the nature, the purpose and the methodology of the research.
* Having signed an informed consent writes before the inclusion in the research.
* Membership or beneficiary of a national insurance scheme

Exclusion Criteria:

* Systematic pathology with neurological appearance
* Psychiatric disorders
* History of psychotic disorders
* History of cranial trauma serious (according to the classification), previous or evolutionary other neurological pathology
* Major protected by the law (supervision or guardianship)
* Loss of liberty by court or administrative order

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2015-07-22 (Actual); Primary Completion 2027-10-22 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Measure of the potential evoked | 2 months
  Measured by electroencephalography and electrocorticography before the beginning of the surgery and before and after the surgical resection

CONTACTS AND LOCATIONS:
Overall Officials: Hugues DUFFAU, Professor, Principal Investigator — Department of neurosurgery, Hospital Gui de Chauliac, Montpellier
Locations (1):
- CHU de Montpellier - Service de neurochirurgie, Montpellier, France

REFERENCES:
- [Background] Rosenwald AG, Krag SS. Lec9 CHO glycosylation mutants are defective in the synthesis of dolichol. J Lipid Res. 1990 Mar;31(3):523-33. PMID 2111370
- [Background] Turpin C, Rossel O, Schlosser-Perrin F, Ng S, Matsumoto R, Mandonnet E, Duffau H, Bonnetblanc F. Shapes of direct cortical responses vs. short-range axono-cortical evoked potentials: The effects of direct electrical stimulation applied to the human brain. Clin Neurophysiol. 2025 Jan;169:91-99. doi: 10.1016/j.clinph.2024.10.016. Epub 2024 Nov 8. PMID 39578190
- [Background] Berger MS, Rostomily RC. Low grade gliomas: functional mapping resection strategies, extent of resection, and outcome. J Neurooncol. 1997 Aug;34(1):85-101. doi: 10.1023/a:1005715405413. PMID 9210055
- [Background] Borchers S, Himmelbach M, Logothetis N, Karnath HO. Direct electrical stimulation of human cortex - the gold standard for mapping brain functions? Nat Rev Neurosci. 2011 Nov 30;13(1):63-70. doi: 10.1038/nrn3140. PMID 22127300
- [Background] DeAngelis LM. Brain tumors. N Engl J Med. 2001 Jan 11;344(2):114-23. doi: 10.1056/NEJM200101113440207. No abstract available. PMID 11150363
- [Background] Duffau H. Lessons from brain mapping in surgery for low-grade glioma: insights into associations between tumour and brain plasticity. Lancet Neurol. 2005 Aug;4(8):476-86. doi: 10.1016/S1474-4422(05)70140-X. PMID 16033690
- [Background] Duffau H, Capelle L, Sichez N, Denvil D, Lopes M, Sichez JP, Bitar A, Fohanno D. Intraoperative mapping of the subcortical language pathways using direct stimulations. An anatomo-functional study. Brain. 2002 Jan;125(Pt 1):199-214. doi: 10.1093/brain/awf016. PMID 11834604
- [Background] Duffau H, Lopes M, Arthuis F, Bitar A, Sichez JP, Van Effenterre R, Capelle L. Contribution of intraoperative electrical stimulations in surgery of low grade gliomas: a comparative study between two series without (1985-96) and with (1996-2003) functional mapping in the same institution. J Neurol Neurosurg Psychiatry. 2005 Jun;76(6):845-51. doi: 10.1136/jnnp.2004.048520. PMID 15897509
- [Background] Duffau H, Sichez JP, Lehericy S. Intraoperative unmasking of brain redundant motor sites during resection of a precentral angioma: evidence using direct cortical stimulation. Ann Neurol. 2000 Jan;47(1):132-5. PMID 10632114
- [Background] Keles GE, Lundin DA, Lamborn KR, Chang EF, Ojemann G, Berger MS. Intraoperative subcortical stimulation mapping for hemispherical perirolandic gliomas located within or adjacent to the descending motor pathways: evaluation of morbidity and assessment of functional outcome in 294 patients. J Neurosurg. 2004 Mar;100(3):369-75. doi: 10.3171/jns.2004.100.3.0369. PMID 15035270
- [Background] Keller CJ, Honey CJ, Megevand P, Entz L, Ulbert I, Mehta AD. Mapping human brain networks with cortico-cortical evoked potentials. Philos Trans R Soc Lond B Biol Sci. 2014 Oct 5;369(1653):20130528. doi: 10.1098/rstb.2013.0528. PMID 25180306
- [Background] Matsumoto R, Nair DR, LaPresto E, Bingaman W, Shibasaki H, Luders HO. Functional connectivity in human cortical motor system: a cortico-cortical evoked potential study. Brain. 2007 Jan;130(Pt 1):181-97. doi: 10.1093/brain/awl257. Epub 2006 Oct 17. PMID 17046857
- [Background] Matsumoto R, Nair DR, LaPresto E, Najm I, Bingaman W, Shibasaki H, Luders HO. Functional connectivity in the human language system: a cortico-cortical evoked potential study. Brain. 2004 Oct;127(Pt 10):2316-30. doi: 10.1093/brain/awh246. Epub 2004 Jul 21. PMID 15269116
- [Background] Szelenyi A, Bello L, Duffau H, Fava E, Feigl GC, Galanda M, Neuloh G, Signorelli F, Sala F; Workgroup for Intraoperative Management in Low-Grade Glioma Surgery within the European Low-Grade Glioma Network. Intraoperative electrical stimulation in awake craniotomy: methodological aspects of current practice. Neurosurg Focus. 2010 Feb;28(2):E7. doi: 10.3171/2009.12.FOCUS09237. PMID 20121442
- [Background] Taphoorn MJ, Klein M. Cognitive deficits in adult patients with brain tumours. Lancet Neurol. 2004 Mar;3(3):159-68. doi: 10.1016/S1474-4422(04)00680-5. PMID 14980531
- [Background] Walker DG, Kaye AH. Low grade glial neoplasms. J Clin Neurosci. 2003 Jan;10(1):1-13. doi: 10.1016/s0967-5868(02)00261-8. No abstract available. PMID 12464515